CLINICAL TRIAL: NCT05129267
Title: Evaluation of Injectable PRF With Vitamin C as an Adjunct to Non-surgical Therapy in the Treatment of Stage II Grade A Periodontitis. A Randomized Controlled Clinical Trial
Brief Title: Evaluation of iPRF With Vitamin C in StageII Grade A Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Abdulhakim Mohamed Sherif, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PER 3- 3- 2
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group B (Active Comparator): Scaling and Root Debridement + iPRF
  Interventions: Other: Group B
- Group C (Active Comparator): Scaling and Root Debridement + iPRF +Vitamin C
  Interventions: Other: Group C
- Group A (No Intervention): Scaling and Root Debridement

INTERVENTIONS:
Other: Group B — Scaling and Root debridement + iPRF
  Arms: Group B
Other: Group C — Scaling and Root debridement + iPRF together with vitamin C
  Arms: Group C

SUMMARY:
Comparing the effect of using vitamin C with injectable PRF as a locally delivered adjunct to scaling and root planing versus scaling and root planing with local delivery of injectable PRF and scaling and root planing alone on the clinical parameters in Stage II Grade A Periodontitis patients.

DETAILED DESCRIPTION:
The conventional approach:

Group 1: Scaling and root planing alone using Gracey curettes and ultrasonic scalers.

Group 2: Scaling and root planing using Gracey curettes and ultrasonic scalers with local delivery of injectable PRF using an insulin syringe with the blunt needle inserted into the bottom of the periodontal pocket through a template to hold the locally delivered injectable PRF.

The intervention approach:

Scaling and root planing using Gracey curettes and ultrasonic scalers with local delivery of vitamin C (250 μM) and injectable PRF, using an insulin syringe with the blunt needle inserted into the bottom of the periodontal pocket through a template to hold the locally delivered vitamin C and injectable PRF for a longer time.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with healthy systemic condition.
2. Adult patients ˃ 18 years old.
3. Patients with Stage II Grade A periodontitis.
4. Patients accept 6-months follow-up period (cooperative patients).
5. Patients provide an informed consent.

Exclusion Criteria:

1. Presence of prosthetic crowns.
2. Extensive restorations.
3. Periodontal therapy within the last 12 months.
4. Having surgical therapy or undergoing orthodontic treatment.
5. Ongoing drug therapy that might have an impact on the clinical signs and symptoms of periodontitis.
6. The use of antibiotics or anti-inflammatory drugs 1 month prior to the procedure and till the end of 6 months of follow-up.
7. Smokers.
8. Pregnant females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-10-03 (Actual); Primary Completion 2022-06-02 (Estimated); Study Completion 2022-06-02 (Estimated)

PRIMARY OUTCOMES:
Bleeding on Probing (BOP) | 3 months
  Gentle probing of the orifice of the gingival crevice. The periodontal probe will be inserted 1 to 2 mm into the gingival sulcus starting at one interproximal area and moving to the other. If bleeding occurs within 10 seconds a positive finding is recorded.

SECONDARY OUTCOMES:
Probing Depth (PD) | 6 months
  Measured from the gingival margin to the bottom of the gingival sulcus. Each tooth will be probed with a light force not exceeding 25 grams at 6 sites.
Clinical Attachment Level (CAL) | 6 months
  Measured from the CEJ to the bottom of the gingival sulcus, or will be calculated as the algebraic sum of gingival recession and PD measurements for each site. Each tooth will be probed with a light force not exceeding 25 grams at six points: (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, and disto-lingual).
Gingival Marginal Level (GML) | 6 months
  Measured from the free gingiva to CEJ.
Plaque Index (PI) | 6 months
  Teeth in each quadrant will be dried with a blast of air, and presence of visible dental plaque will be recorded with scores 0, 1, 2, 3.
Intraoral Radiographs | 6 months
  A customized X-ray positioning stent will be fabricated to allow easy and accurate radiographing and retain the plastic film holder in the paralleling radiographic technique.
Post-Operative Pain | 48 hours
  Visual Analogue Scale (VAS) with numbers from 0 to 10 ('no pain' to 'worst pain imaginable') measured daily for the first 2 days postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medecine-CU, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sherif MA, Anter E, Graetz C, El-Sayed KF. Injectable platelet-rich fibrin with vitamin C as an adjunct to non-surgical periodontal therapy in the treatment of stage-II periodontitis: a randomized controlled clinical trial. BMC Oral Health. 2025 May 23;25(1):772. doi: 10.1186/s12903-025-06115-x. PMID 40410805